CLINICAL TRIAL: NCT04296123
Title: Psychometric Properties of Four Step Tests and Effects of Step Training in Reducing Falls on Older Adults with Dementia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, Dr. Wayne Chan, Assistant Professor, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: WC-20200302002
Record Dates: First submitted 2020-03-02; First posted 2020-03-05 (Actual); Last update posted 2024-10-04 (Actual); Status verified 2024-10

CONDITIONS: Dementia
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental)
  Interventions: Behavioral: Step training
- Control (No Intervention)

INTERVENTIONS:
Behavioral: Step training — A 12-week step training consisting of two 30-minute training session per week. The participants will be instructed to stand upright and step on different targets on a plastic mat repeatedly.
  Arms: Intervention

SUMMARY:
Abstract:

Objectives: (i) To investigate the test-retest and inter-rater reliability, construct and known-group validity of four independent step tests in older adults with mild to moderate dementia (Phase 1); and (ii) the feasibility and effects of a 12-week step training on the step performance, physical and functional outcomes in this population (Phase 2).

Design and subjects: Older adults who have mild to moderate dementia, and able to walk independently without walking aids, with stick or quadripod will be recruited to participate in this study. Participants will perform four step tests, including Four Square Step Test (FSST), Choice Stepping Reaction Time Test (CSRTT), Maximum Step Length Test (MSLT) and Alternate Step Test (AST) on three separate testing occasions conducted by two independent raters at the baseline (Phase 1).

The participants will then join either an intervention or control group. Those in the intervention group will receive a 12-week step training, while the control group will receive usual care. The stepping performance using the step tests validated in Phase 1, cognitive and functional outcomes and prospective falls will be compared between the intervention and control groups at 12 and 24 weeks (Phase 2).

Interventions: The step training consists of two 30-minute training sessions per week. The participants will receive an individualized, progressive training that is tailored to their stepping ability and cognitive function.

Main outcome measures: Stepping performance using the four step tests, 2-minute walk test, 10-meter walk test, 30-second sit to stand test, Berg Balance Scale, Montreal Cognitive Assessment and prospective falls at 12 and 24 weeks.

Expected results: (i) The four step tests are reliable in older adults with mild to moderate dementia, and the findings of the step tests are moderately associated with the functional outcomes, and (ii) the participants in the intervention group will have better stepping performance, better functional outcomes and fewer falls compared with the control group at 12 weeks, and the effects will sustain at 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

* 65 years or above
* able to walk independently without walking aid, with stick or quadripod
* clinical diagnosis of dementia

Exclusion Criteria:

* unstable cardiac or pulmonary conditions
* acute musculoskeletal or severe neurological conditions affecting stepping performances
* severe hearing or visual impairment limiting communication
* severe cognitive impairment
* recent hospitalization in the past 30 days

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 47 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2024-03-31 (Actual); Study Completion 2024-03-31 (Actual)

PRIMARY OUTCOMES:
Four Square Step Test | 12 weeks
Four Square Step Test | 24 weeks
Choice Stepping Reaction Time Test | 12 weeks
Choice Stepping Reaction Time Test | 24 weeks
Maximum Step Length Test | 12 weeks
Maximum Step Length Test | 24 weeks
Alternate Step Test | 12 weeks
Alternate Step Test | 24 weeks

SECONDARY OUTCOMES:
10-meter walk test | 0, 12 and 24 weeks
2-minute walk test | 0, 12 and 24 weeks
30-second sit to stand test | 0, 12 and 24 weeks
Berg balance scale | 0, 12 and 24 weeks
  The score ranges from 0-56. A higher score indicates better balance control
Number of falls | 0, 12 and 24 weeks
Montreal Cognitive Assessment | 0, 12 and 24 weeks
  The score ranges from 0-30. A higher score indicates better global cognitive function

CONTACTS AND LOCATIONS:
Overall Officials: Wayne Chan, PhD, Principal Investigator — The Hong Kong Polytechnic University
Locations (1):
- The Hong Kong Polytechnic University, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Chan WLS, Tsang SMH, Ho LYW. Reliability and Validity of Four Step Tests in Older Adults With Dementia. Int J Geriatr Psychiatry. 2024 Dec;39(12):e70021. doi: 10.1002/gps.70021. PMID 39608824